CLINICAL TRIAL: NCT03395418
Title: Evaluation of the Right Use of Inhaled Therapeutics Prescribed in Asthma and COPD in Adults
Brief Title: Evaluation of the Right Use of Inhaled Therapeutics
Acronym: ARGOS
Status: Completed | Type: Observational
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02599-44
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: COPD Asthma
Keywords: COPD; Asthma; Inhaled Therapeutics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma and COPD have a significant impact on public health, affecting about 8 million people in France and generating health care costs of 5.5 billion euros, almost 50% of which are dedicated to long-term treatments are essentially inhaled therapies.

The good control of the disease depends on the patient's compliance, but also on the proper use of the devices used for the administration of inhaled drugs under penalty of the degradation of the control of the disease with major medical and medico-economic consequences.

Thus, education of these patients in the use of devices must be an integral part of medical care. It comes up against the complexity of the therapeutic arsenal on the one hand and on the other hand with its time-consuming nature: this makes it incompatible with a realization in consultation.

The "ARGOS" process is a telemonitoring project for the support of therapeutic education, consisting in setting up a concrete and real-time relay between prescribers and patients for the education of inhaled therapeutics.

Its objective is to provide the answer to what is currently an "unmet need" in the management of asthma and COPD, with the prospect of a positive impact on the observance of these treatments and by consequently their clinical and economic efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed in Pneumology for asthma or COPD with a prescription for long-term inhaled therapies AND a home health provider (who monitors either home oxygen and / or respiratory equipment)
* The patient must have a means of telephone communication in order to be able to be contacted by a provider, an H2AD permanence or a doctor
* Patient having given his agreement after having been informed in writing of the purpose and the data collected during this study
* Age ≥ 18 years
* Beneficiary of a social security scheme

Exclusion Criteria:

* Refusal of the patient
* Patient not understanding French
* Absence of home health provider
* Absence of means of telephone communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in pneumology for asthma or COPD who have:
  * a prescription for long-term inhaled therapeutics
  * also a home health provider (either for long-term oxygen or for a CPAP, NIV ...)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of exploitable films | Day 1 to day 7
  Ratio between the number of exploitable films and the number of films arriving at the telemedicine platform.

CONTACTS AND LOCATIONS:
Locations (1):
- ANTADIR, Paris, France